CLINICAL TRIAL: NCT07016308
Title: Effects of Low-Flow Desflurane and Sevoflurane Anesthesia on Physiological Parameters and Recovery Process
Brief Title: Low-Flow Desflurane vs Sevoflurane: Impact on Physiology and Recoveryand Recovery Profiles in Adult ENT Surgery
Acronym: LoFADS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Veli Fahri Pehlivan, Assistant Professor, Harran University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ceren
Record Dates: First submitted 2025-05-30; First posted 2025-06-11 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Anesthesia, General
Keywords: Sevoflurane; Desflurane; Low-flow anesthesia
MeSH Terms: interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive either low-flow sevoflurane or low-flow desflurane anesthesia.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Both participants and outcome assessors will be blinded to group allocation. Anesthesia providers will use coded gas assignments to ensure blinding during the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane Low-Flow Anesthesia (Experimental): Participants in this group will receive general anesthesia using sevoflurane administered under low-flow conditions. After standard induction and intubation, sevoflurane will be maintained at 2-3% (0.8-1 MAC) with a fresh gas flow of 1 L/min (50% oxygen / 50% air). Vital signs and arterial blood gases will be monitored, and recovery parameters such as time to spontaneous breathing, extubation, and verbal response will be recorded.
  Interventions: Drug: Sevoflurane; Drug: Desflurane
- Desflurane Low-Flow Anesthesia (Active Comparator): Participants in this group will receive general anesthesia using desflurane administered under low-flow conditions. After standard induction and intubation, desflurane will be maintained at 4-6% (0.8-1 MAC) with a fresh gas flow of 1 L/min (50% oxygen / 50% air). Hemodynamic and respiratory parameters as well as arterial blood gases and recovery times will be evaluated and compared to the sevoflurane group.
  Interventions: Drug: Sevoflurane; Drug: Desflurane

INTERVENTIONS:
Drug: Sevoflurane — Sevoflurane will be administered via inhalation under low-flow anesthesia conditions. The concentration will be maintained at 2-3% (0.8-1 MAC) with a fresh gas flow of 1 L/min (50% oxygen and 50% air) after induction. Used in Group S (Sevoflurane Low-Flow Anesthesia Arm).
Drug: Desflurane — Desflurane will be administered via inhalation under low-flow anesthesia conditions. The concentration will be maintained at 4-6% (0.8-1 MAC) with a fresh gas flow of 1 L/min (50% oxygen and 50% air) after induction. Used in Group D (Desflurane Low-Flow Anesthesia Arm).
  Other Names: Suprane

SUMMARY:
This randomized, double-blind, controlled clinical trial aims to compare the effects of low-flow sevoflurane and desflurane anesthesia on physiological parameters and recovery profiles in adult patients undergoing ENT surgeries. The primary outcomes include heart rate, mean arterial pressure, peripheral oxygen saturation, end-tidal CO₂, and arterial blood gas values. Secondary outcomes involve time to spontaneous respiration, extubation, and response to verbal commands.

DETAILED DESCRIPTION:
This prospective study investigates the clinical effects of low-flow anesthesia using two commonly utilized volatile agents, sevoflurane and desflurane, in adult patients undergoing elective ENT surgeries, specifically rhinoplasty, mastoidectomy, and tympanoplasty. A total of 40 ASA I-II patients, aged 18-65, will be randomly assigned into two groups: Group S (sevoflurane) and Group D (desflurane).

All participants will undergo general anesthesia with endotracheal intubation. After 2 minutes of preoxygenation with 100% oxygen at 10 L/min, anesthesia will be induced and maintained with the assigned volatile agent under low-flow settings (1 L/min, 50% O₂-50% air). Hemodynamic and respiratory parameters (HR, MAP, SpO₂, EtCO₂) will be recorded at predefined time points, along with arterial blood gas analysis (pH, pCO₂, pO₂, COHb).

Recovery times including return of spontaneous respiration, extubation, and verbal response will be documented. This study aims to provide clinical evidence on the optimal anesthetic choice under low-flow conditions, supporting safer, more efficient, and environmentally conscious anesthesia practices.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 65 years
* Classified as ASA physical status I or II
* Scheduled to undergo elective ENT surgery (rhinoplasty, mastoidectomy, or tympanoplasty)
* Requiring general anesthesia with endotracheal intubation
* Providing written informed consent

Exclusion Criteria:

* ASA physical status III or higher
* History of malignant hyperthermia or delayed emergence from anesthesia
* Morbid obesity (BMI ≥ 35)
* Coronary artery disease, congestive heart failure, COPD, liver or kidney disease
* Pregnancy or breastfeeding
* Allergy to halogenated anesthetics
* Respiratory pathology
* Substance or alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in Heart Rate During Surgery | From preoperative baseline to 120 minutes after anesthesia induction
  Heart rate (HR) will be measured at baseline, post-intubation, and at 15, 30, 45, 60, and 120 minutes after anesthesia induction.
Change in Mean Arterial Pressure During Surgery | From preoperative baseline to 120 minutes after induction
  Mean arterial pressure (MAP) will be recorded at the same predefined time intervals during surgery.
Change in End-Tidal CO₂ | From preoperative baseline to 120 minutes after induction
  End-tidal carbon dioxide (EtCO₂) levels will be monitored during surgery at specified intervals.
Change in Peripheral Oxygen Saturation | From preoperative baseline to 120 minutes after induction
  Peripheral oxygen saturation (SpO₂) will be measured at baseline, post-intubation, and intraoperative time points.

SECONDARY OUTCOMES:
Change in Arterial pH | Preoperative, intraoperative (60 and 120 min), end of surgery
  Arterial blood gas samples will be analyzed for pH at baseline, 60 and 120 minutes, and at end of surgery.
Post-Anesthesia Recovery Times | From end of surgery until recovery (within approx. 30 minutes)
  Time to return of spontaneous respiration, time to extubation, and time to follow verbal commands will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Basak Pehlivan, Asoc Prof. Dr, Principal Investigator — Harran University
Locations (1):
- Veli Fahri Pehlivan, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No